CLINICAL TRIAL: NCT02946281
Title: Do Cardiac Health: Advanced New Generation Ecosystem
Acronym: Do CHANGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elisabeth-TweeSteden Ziekenhuis (Other)
Collaborators: Eindhoven University of Technology (Other); Smart Homes (Unknown); Badalona Serveis Assistencials (Other); Docobo Ltd. (Industry); Do Something Different (Other); Fundació Eurecat (Other); ONMI (Unknown); ITRII (Unknown); Buddhist Tzu Chi General Hospital (Other); European Commission (Other)
Responsible Party: Principal Investigator, Jos Widdershoven, Prof. Dr., Elisabeth-TweeSteden Ziekenhuis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: L0264.2016
Record Dates: First submitted 2016-07-07; First posted 2016-10-27 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Lifestyle
Keywords: self-management; health behavior; cardiac disease; habits; lifestyle
MeSH Terms: conditions — Health Behavior; Heart Diseases; Habits

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: Do CHANGE
- Care as usual (No Intervention)

INTERVENTIONS:
Behavioral: Do CHANGE — The intervention aims to increase behavioral flexibility and change patients' (unhealthy) lifestyle. At the same time the intervention should increase patient self-management and improve the patient reported outcomes (e.g. quality of life, anxiety, depression).
  Other Names: Do Something Different; Docobo Care Portal; Moves app; Blood pressure monitor UA -767 Plus
  Arms: Intervention

SUMMARY:
The primary objective of Do CHANGE is to develop a health ecosystem for integrated disease management of citizens with high blood pressure and patients with ischemic heart disease or heart failure. The system will give them access to a set of personalized health services in a near real-time fashion. This disruptive system will incorporate the behaviour change methods, such as "Do Something Different", in conjunction with new innovative wearable/portable tools that can monitor behaviour and clinical parameters in normal living situations.

DETAILED DESCRIPTION:
Patients enrolled for participation will be randomly assigned to the intervention or 'care as usual' group (1:1). Patients assigned to the intervention group will receive a 3 month intervention aiming to enhance self-management and lifestyle.

The intervention will consist out 4 components.

1. Behavioral prompts (Do's) from the Do Something Different Programme The Do Something Different Program has previously been developed and evaluated (ref). For the current study, the programme has been adapted to the population of interest (CAD, HF, and HT patients) together with behavioural experts and cardiologists. The program aims to change behavioural habits and increase flexibility and subsequently change habits associated with an unhealthy lifestyle and distress, which are both found to be associated with hypertension and cardiovascular risks. The program has been developed with input from cardiologists , psychologists, and patients. 'Typical' other behavioural risks besides hypertension have been identified and are addressed within the program. To further adapt the program to patient' needs, all patient, prior to starting the program, will be assessed regarding their own functioning, distress, and personality such that the Do's will match their personal habits and challenge them to change.

   After assessing patients personality profile the intervention will be provided for 11 weeks. Patients will receive a total of 32 Do's / messages during this period. The Do's will be matched to their personal profile.
2. Care-Portal All patients who are randomized to the intervention group will also receive a Care-Portal (Docobo Ltd.) which will be installed at their home. The Care-Portal will be used to gather ECG data and blood pressure on a daily basis. The Care-Portal will send the physiological data directly to the cardiologist who will be able to access those via an online platform and contact the patient if necessary.

   In addition, patients will receive their Do's trough the care-portal. The Care-Portal is a CE-marked device that has previously been successfully used and implemented to support patients with chronic conditions.
3. Blood pressure monitor All patients in the intervention group will receive the digital blood pressure monitor 'UA -767 Plus' which is a CE-marked device for clinical use. Patients will be asked to measure their blood pressure on a daily basis and record the values through the care-portal.
4. Moves App For the future study within the Do CHANGE project, the Do Something Different programme wants to focus on providing 'Contextual Do's' where patients will receive behavioural prompts at the moment that the behaviour takes place. In order to reach this goal getting more insight in patients behavioral patters is of utmost importance. Hence, that data will be gathered within this current study as one of the exploratory objectives using GPS data. This will give more insights and will be used as input for future study. All patients participating in the intervention will be provided with the 'Moves' app that will log their activities anonymously. This information will automatically be available for research purposes only. Patients will not receive any push messages from that app or any feedback.

"Moves" is an automatic diary of patients life. The daily storyline and maps show where, when, and how much a person moves. The application automatically records any walking, cycling, and running that is done. The app is always active in the background, so there's no need to start and stop it. Just keep the phone in the pocket or a bag. The app consumes battery power, so nightly charging is recommended. With typical phone use, a smartphone running Moves should have enough battery power to last all day. The optional Battery Saving Mode in Moves for iPhone saves up to 40% of battery.

The Moves API can be used to build new apps, integrate with an existing service and visualise data. The API is designed for apps and services that have a server component. Individual users need to give permission to access data. However, providing any kind of personal information is optional, data collection can be done anonymously as well. Moves uses OAuth 2.0 for authentication and authorization and the actual authorization happens in the Moves app.

During this study the API can be used to collect location based data from participants. This data will be used to develop the location based responsive Do program. During the study participants will not receive feedback from the application. In the settings all notifications can be turned off. Besides, the app can be used without setting goals and accounts. The only thing a participant is asked is to install the app and fill in a unique code for data collection. Participants who do not use a smartphone or are not able to install the app do not have to use it.

ELIGIBILITY:
Inclusion Criteria:

* age 18-75 years
* diagnosed with CAD, HF or HT
* having at least two of the following risk factors: smoking, positive family history, increased cholesterol, diabetes, sedentary lifestyle, psychosocial risk factors.
* Patients should also have access to the Internet and have a smartphone (and sufficient knowledge on using personal computer or smartphone)
* Patients should have sufficient knowledge of the countries' native language.
* Additional inclusion criteria for HF patients only is to have a left ejection fraction of ≤35% and experience HF symptoms (e.g. shortness of breath, chest pain, exhaustion).

Exclusion Criteria:

* significant cognitive impairments (e.g. dementia)
* patients who are on the waiting list for heart transplantation
* life expectancy <1 year
* life threatening comorbidities (e.g. cancers)
* history of psychiatric illness other than anxiety/depression
* patients who do not have access to internet
* patients with insufficient knowledge of the local pilot language (Dutch, Chinese and Catalonian).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2016-12-19 (Actual); Primary Completion 2017-12-22 (Actual); Study Completion 2017-12-22 (Actual)

PRIMARY OUTCOMES:
Lifestyle | 0-6 months
  The Health Promoting Lifestyle Questionnaire (HPLP-II) will be administered to evaluate whether patients' subjective perception of lifestyle change has changed.
Behavioural flexibility | 6 months
  Whether the patients' behavioural flexibility (having a bigger behavioural repertoire which makes it easier to perform alternative behaviours) has increased and thus whether behaviour change (as conceptualized by Do Something Different program) has occurred will be assessed using purpose designed questions by the Do Something Different program.
Quality of life | 6 months
  Changes in quality of life will be assessed using the WHOQOL-Bref questionnaire. As this is a widely used instrument it will allow the integration of data from different partners.

SECONDARY OUTCOMES:
Usability, acceptance, satisfaction with intervention / tools | 3 months
  Unified Theory of Acceptance and Use of Technology (UTAUT2) questionnaire will be used to assess the usability, acceptance, and satisfaction of the care portal.
Cost-effectiveness | 6 months
  Whether the intervention arm will be cost-effective as compared to the care as usual will be evaluated using the EQ-5D questionnaire. It could be expected that the intervention arm will experience a lower disease burden and be less likely to use additional health care resources.

OTHER OUTCOMES:
Depression | 6 months
  The Patient Health Questionnaire (PHQ-9) will be use to assess depression within the sample.
Anxiety | 6 months
  The Generalized Anxiety Disorder (GAD-7) questionnaire will be used to assess the levels of anxiety.
Lifestyle data sensor generated | 3 months
  Patients' physical activity will be monitored (pedometer / active minutes per day) and evaluated by comparing their daily amount of steps / activity pre and post intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Jos Widdershoven, Prof. dr., Principal Investigator — Elisabeth-TweeSteden Ziekenhuis
Locations (2):
- Elisabeth-TweeSteden Hospital, Tilburg, North Brabant, Netherlands
- Badalona Serveis Assistencials, Badalona, Spain

REFERENCES:
- [Derived] Habibovic M, Piera-Jimenez J, Wetzels M, Widdershoven JWGM, Soedamah-Muthu SS. Associations between behavioral flexibility and health behavior in cardiac patients in the Do CHANGE trials. Health Psychol. 2022 Oct;41(10):710-718. doi: 10.1037/hea0001151. Epub 2022 May 16. PMID 35575702
- [Derived] Broers ER, Kop WJ, Denollet J, Widdershoven J, Wetzels M, Ayoola I, Piera-Jimenez J, Habibovic M. A Personalized eHealth Intervention for Lifestyle Changes in Patients With Cardiovascular Disease: Randomized Controlled Trial. J Med Internet Res. 2020 May 22;22(5):e14570. doi: 10.2196/14570. PMID 32441658